CLINICAL TRIAL: NCT03674229
Title: Using Patient Navigators to Facilitate Weight Management Among Adults
Brief Title: Patients Navigators in Facilitating Weight Management in Obese Participants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-0255; NCI-2018-01819 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2018-09-10; First posted 2018-09-17 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Health Status Unknown; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (information about weight management programs) (Active Comparator): Participants receive information about commercially-available weight management programs and encouragement to participate in one of the programs for 6 months.
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration
- Group II (information, call from patient navigator) (Experimental): Participants receive information about commercially-available weight management programs encouragement to participate in one of the programs for 6 months. Participants also receive 6 phone calls over 20-30 minutes each from an assigned patient navigator for 6 months.
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Informational Intervention — Receive information about weight management programs
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive phone calls from an assigned patient navigator
  Arms: Group II (information, call from patient navigator)

SUMMARY:
This trial studies the effectiveness of patient navigators in facilitating weight management in obese participants. Health coaches or patient navigators may help more participants take part in weight management programs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effectiveness of patient navigators to increase enrollment in evidence-based weight management programs.

SECONDARY OBJECTIVES:

I. To evaluate the effectiveness of patient navigators to increase overall attendance or use of evidence-based weight management programs.

II. To evaluate the effectiveness of patient navigators to promoting and facilitating positive health behavior change: increased physical activity; improved diet; and weight loss.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants receive information about commercially-available weight management programs and encouragement to participate in one of the programs for 6 months.

GROUP II: Participants receive information about commercially-available weight management programs encouragement to participate in one of the programs for 6 months. Participants also receive 6 phone calls over 20-30 minutes each from an assigned patient navigator for 6 months.

After completion of the study, participants are followed up at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Are referred by a University of Texas (UT) health care provider
* Have a body mass index (BMI) greater than or equal to 30 and less than or equal to 45 kg/m^2
* Are able to read and speak English
* Have a working telephone number and address where materials can be mailed
* Able to engage in moderate intensity physical activity as determined by the Physical Activity Readiness Questionnaire (PAR-Q)
* Internet access at home or other location (e.g., work, church, library, community center, etc.)

Exclusion Criteria:

* Another person in the same household already enrolled in the proposed intervention
* Pregnant or thinking about becoming pregnant during the study period
* Are already involved in another weight loss program
* Participated in a weight loss, exercise, or dietary modification program in the previous 6 months
* Involuntary or voluntary weight loss of greater than or equal to 5% body weight in the previous 6 months
* Are currently using weight loss medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in participant enrollment in evidence-based weight management programs | Up to 6 months
  We will compare differences in the proportion of self-reported enrollment in any program between intervention and control groups.

SECONDARY OUTCOMES:
Participant attendance or use of evidence-based weight management programs | Up to 6 months
  Attendance is a continuous variable and is defined as the total number of self-reported sessions attended or used by each participant.
Positive change in physical activity | Baseline up to 6 months
  Accelerometer data will provide an objective assessment of physical activity (PA) We will calculate minutes of PA per week and meeting recommendations (yes/no).
Measurement of fruit and vegetable consumption | Baseline up to 6 months
  Fruit and vegetable consumption (i.e., # servings per day) will be measured using the 24 hour recall. Finally, objective measure of weight will be captured at each data collection time point.
Objectively measured weight change. | Baseline up to 6 months
  Change in body weight from baseline will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna McNeill, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Heredia NI, Fernandez ME, van den Berg AE, Durand CP, Kohl HW, Reininger BM, Hwang KO, McNeill LH. Coaction Between Physical Activity and Fruit and Vegetable Intake in Racially Diverse, Obese Adults. Am J Health Promot. 2020 Mar;34(3):238-246. doi: 10.1177/0890117119884479. Epub 2019 Nov 13. PMID 31722544
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org